CLINICAL TRIAL: NCT03903224
Title: Effect of Combined Modified Pectoralis and Transversus Plane Blocks Versus Erector Spinae Block on Postoperative Analgesia Following Modified Radical Mastectomy
Brief Title: Combined PECS II and Transversus Plane Blocks Versus Erector Spinae Block in Modified Radical Mastectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Bakri, Professor doctor of anaesthesia and ICU Faculty of Medicine - Assiut University, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Analgesia in breast surgey
Record Dates: First submitted 2019-03-29; First posted 2019-04-04 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Breast Cancer; Acute Postoperative Pain
Keywords: Breast Cancer; Regional Anaesthesia; Morphine Consumption
MeSH Terms: conditions — Breast Neoplasms; Pain, Postoperative | interventions — thiamine triphosphorate

STUDY DESIGN:
Who Masked: Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Combined PECS II and TTP blocks (PT) (Active Comparator): Modified Pectoralis block (PECS II) : Using ultrasound we proceed to inject 10 ml of bupivacaine 0.25% between the pectoral muscles and 10 ml under Pmm above the serratus muscle.
  Transversus Thoracic Plane block : 10 mL bupivacaine (0.25%) is injected between the transversus thoracic muscle and the internal intercostal muscle between the third and fourth left ribs connecting at the sternum.
  Interventions: Procedure: Combined Modified Pectoralis and Transversus Plane Blocks
- Erector Spinae Block (E) (Active Comparator): Using ultrasound an echogenic 22-G block needle is inserted in-plane in a cranial-to-caudal direction until contact is made with the T5 transverse process. A total of 30 bupivacaine 0.25% is then injected while seeing the fluid lifting the erector spinae muscle off.
  Interventions: Procedure: Erector Spinae block

INTERVENTIONS:
Procedure: Combined Modified Pectoralis and Transversus Plane Blocks — Modified pectoralis nerve block (Pecs II) aims to block at least the pectoral nerves, the intercostobrachial, intercostals III-IV-V-VI. This will cover dermatomes T2, T3 and T4. The probe is positioned under the lateral third of the clavicle .After locating the subclavian muscle, the axillary artery and the axillary vein we move the probe distally towards the axilla, until the pectoralis minor is identified. We start counting the ribs , from r1 under the axillary artery, we move distally and laterally until the lateral border of pectoralis minor is reached. The serratus anterior muscle which covers r2, r3, r4 is the point of entrance into the axilla.
  Blocking of multiple anterior branches of intercostal nerves (Th2-6) using a transversus thoracic muscle plane (TTP) block is used as an additive to pecs II to cover the internal mammary region
  Other Names: PECS II and TTP
  Arms: Combined PECS II and TTP blocks (PT)
Procedure: Erector Spinae block — The patient is placed in a sitting position and The T5 spinous process is located by palpating and counting down from the C7 spinous process. Under complete aseptic conditions a linear ultrasound probe is then placed in a transverse orientation at the level of the T5 transverse process. The tip of the transverse process is centred on the ultrasound screen and the probe is then rotated into a longitudinal orientation to produce a parasagittal view. From T1 to T5 the erector spinae, rhomboid major and trapezius muscles are visible posterior and superficial to the transverse processes.
  Arms: Erector Spinae Block (E)

SUMMARY:
The aim of this study is to compare the total morphine consumption in the first 24 hour postoperative between combined modified pectoralis block (PECS II) and transversus plane block versus erector spinae block in modified radical mastectomy.

DETAILED DESCRIPTION:
Breast cancer is the most common malignancy in women in the United States and is second only to lung cancer as a cause of cancer death. Breast surgery is commonly performed as a part of the management of breast cancer, is associated with considerable acute postoperative pain. Ultrasound guided Regional anesthesia is recommended to be a part of multimodal analgesia in order to manage the acute post-operative pain. New techniques are proposed to give adequate control of postoperative analgesia with less opioid needs in the first day postoperative. They include pectoralis nerve modified pectoralis, and erector spinae blocks.

The investigators will compare Modified pectoralis nerve block (Pecs II) plus transversus thoracic muscle plane (TTP) block versus Erector spinae block on morphine consumption during first 24 h following modified radical mastectomy.

ELIGIBILITY:
Inclusion Criteria:

* Age 18: 60 years old
* ASA (American Society of Anesthesiologists) physical status I II
* Female patients scheduled for modified radical mastectomy

Exclusion Criteria:

* Patient refusal or inability to give informed consent
* Subjects with a medical contraindication to regional anesthesia , such as coagulopathy, local infection or an allergy to local anesthetic
* Body mass index (BMI) >35
* Presence of psychiatric diseases
* History of chronic chest wall pain or neuropathic disorders
* Alcohol or drug abuse
* Severe chest wall deformities

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2021-02-08 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
The total morphine consumption postoperative (mg) | The first 24 hours postoperative.
  Morphine consumption in mg

SECONDARY OUTCOMES:
Postoperative pain score by Verbal numeric rating scale | 0, 2, 4, 8, 12, 24 hours postoperatively.
  Verbal numeric rating scale (VNRS) for postoperative pain monitoring using 11-point where zero equals no pain and 10 equals the worst pain imaginable.
Time to first request analgesia postoperative (min) | The first 24 hours postoperatively
  Time from postoperative period to time of first analgesic request in minutes
Postoperative level of IL6 (interleukin 6) (pg/mL) | Two blood samples will be withdrawn from the patient. The first one is immediately preoperative and the second one after 24 hours postoperative
  Preoperative baseline and postoperative levels of IL6 will be measured (pg/mL)
Arterial blood gas: Arterial blood gas: Arterial blood gases | Before surgery and 24 hours postoperative.
  Oxygen (mmHg) and carbon dioxide (mmHg)

CONTACTS AND LOCATIONS:
Overall Officials: Eman A Ismail, A Lectuer, Study Director — Assiut University
Locations (1):
- Assiut University Hospital, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol

REFERENCES:
- [Background] Gurkan Y, Aksu C, Kus A, Yorukoglu UH, Kilic CT. Ultrasound guided erector spinae plane block reduces postoperative opioid consumption following breast surgery: A randomized controlled study. J Clin Anesth. 2018 Nov;50:65-68. doi: 10.1016/j.jclinane.2018.06.033. Epub 2018 Jul 2. PMID 29980005